CLINICAL TRIAL: NCT01250652
Title: Efficacy and Safety of 20 mg Levocetirizine and 15 mg Levocetirizine + 50 mg Bed-Time Hydroxyzine in Severe Chronic Urticaria in Adults: a Pilot, Randomized, Double-blind, Cross-over and Parallel, Active-controlled, Single-centre Study
Brief Title: Levocetirizine Plus Bed-Time Hydroxyzine in the Management of Corticodependent Chronic Urticaria Versus Levocetirizine Alone in High Doses
Acronym: LevoHydroxy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Association Asthma, Bulgaria (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Principal Investigator, Prof. Todor Popov, Prof. Todor Popov, Association Asthma, Bulgaria
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 67LH13102010
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Urticaria
Keywords: Chronic urticaria; Urticaria; Antihistamine
MeSH Terms: conditions — Chronic Urticaria; Urticaria | interventions — levocetirizine; Hydroxyzine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levocetirizine (Active Comparator): 24 patients will received 20 mg Levocetirizine daily
  Interventions: Drug: Levocetirizine
- Levocetirizine plus Hydroxyzine (Experimental): 24 patient will receive 15 mg Levocetirizine plus 50 mg Hydroxyzine at bad time for 5 days
  Interventions: Drug: Levocetirizine plus Hydroxyzine

INTERVENTIONS:
Drug: Levocetirizine — 20 mg levocetirizine for 5 days
  Other Names: Xyzal
  Arms: Levocetirizine
Drug: Levocetirizine plus Hydroxyzine — 24 patient will receive 15 mg Levocetirizine plus 50 mg Hydroxyzine at bad time for 5 days
  Other Names: Xyzal plus Atarax
  Arms: Levocetirizine plus Hydroxyzine

SUMMARY:
Allen Kaplan is a prominent American allergist with the reputation of leader in the field of chronic urticaria. He advocates treatment with first generation hydroxyzine, which he considers at least as effective as modern second generation H1-blockers in suppressing the symptoms of difficult-to-treat / systemic-steroid-dependant cases of chronic urticaria. He further speculates that hydroxyzine may have the advantage to better suppress itch and improve nighttime sleep. This has prompted many practitioners around the world to believe that adding hydroxyzine to the treatment regimen at bed time at night may be beneficial to patients. At the same time European guidelines indicate modern second generation H1-blockers in higher than conventional doses as drugs of choice for such cases. However, there is no evidence from clinical trials addressing this controversy. The investigators' previous studies suggest that levocetirizine at quadruple doses may be beneficial in difficult to treat urticaria by reducing lesions and itch, improving quality of life and night time sleep, while not causing day time somnolence. First generation H1-receptor antagonists and hydroxyzine among them are known to penetrate the blood / brain barrier and to cause sedation. The question stays whether this sedation is beneficial to the subjects with chronic urticaria at night, whether it has any hang-over unwanted effects the following day and whether this has any influence on the overall urticaria-specific quality of life.

DETAILED DESCRIPTION:
Study design:

The study will involve two distinct parts (flow chart):

1. In-hospital assessment of effectiveness and tolerability of 10 & 20 mg levocetirizine vs. 100 & 200 mg hydroxyzine in subjects to be weaned off corticosteroid treatment.
2. Subsequent ambulatory treatment of the same patients with 20 mg levocetirizine alone and 15 mg levocetirizine + 50 hydroxyzine at night

Protocol description Patients with chronic urticaria treated with systemic steroids are traditionally admitted to the Clinic of Allergy and Asthma in Sofia to try to wean them off this class of drugs. Hospitalized patients will be invited to take part in the study and will sign an informed consent. They will be assessed by standard questionnaire and by objective assessment of the urticarial lesions, QoLQ will be filled in, discomfort due to urticaria, day time somnolence and night time sleep quality will be assessed on a visual analogue scale. Systemic steroids will be withheld and patients would be given 10 mg levocetirizine on Days 1 & 2; after a new assessment of quality of night time sleep and day time somnolence, 100 mg hydroxyzine will be given on Days 3 & 4. The cycle will be repeated on Days 5 & 6 and Days 7 & 8 with 20 mg levocetirizine and 200 hydroxyzine respectively. At this point patients will be discharged and randomized to two treatment arms: levocetirizine 20 mg per day and levocetirizine 15 mg + hydroxyzine 50 mg as evening dose for 5 days. Diaries will be given to patients for assessment of daily SS, day time somnolence score, quality of night time sleep, facial tissue swelling, rescue medication with oral prednisolone, adverse events, intake of any other medications. After 5 days the patients from arm 1 and 2 will be crossed over to the alternative treatment. QoLQ questionnaire will be filled out at onset, at cross over (day 5) and at the end of the 10 day treatment period. On completion of the study subjects will be asked to state there preference for one treatment or the other.

ELIGIBILITY:
Inclusion Criteria:

* 24 randomized patients of either sex,
* ≥18 years of age.
* Included patients should have at least a 6-week documented history of urticaria with intake of 15-30 mg Prednisolon.

Exclusion Criteria:

* Patients with physically induced urticarias;
* pregnancy and lactation;
* any chronic disease requiring daily other drug treatment including, antihypertensives, antipsychotics and antidepressants;
* other skin disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-03; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Urticaria specific quality of life | 1 year
  The primary objective of the study is to compare the effect on urticaria specific quality of life of two regimens: levocetirizine 20 mg per day (4x1 tablets) vs. levocetirizine 15 mg (3x1 tablets) + hydroxyzine 50 mg (2 tablets) before night time sleep.

SECONDARY OUTCOMES:
Effect of the two regimens on urticaria symptoms | 1 year
  To compare the effect of the two regimens on urticaria symptoms (number of wheals, pruritus severity
Effect on night time sleep | 1 year
  To compare the effect of the two regimens on the quality of night time sleep
Effect on day time somnolence | 1 year
  To compare the effect of the two regimens on the day time somnolence.
The effect on blood eosinophil numbers, Na+, K+, ALAT, ASAT, ECG | 1 year
  To document the effect of treatment with higher doses of levocetirizine or hydroxyzine on blood eosinophil numbers, Na+(sodium ion), K+(potassium ion), ALAT (Alanine transaminase), AST (Aspartate transaminase), ECG (Electrocardiogram)
To assess adverse events | 1 year
  To investigate safety by assessing the nature, incidence and severity of adverse events within the treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Todor A Popov, MD, PhD, Principal Investigator — Professor of Allergology
Locations (1):
- Medical University Sofia, Department of Allergology, Sofia, Bulgaria

REFERENCES:
- [Background] Kaplan AP. Chronic urticaria: pathogenesis and treatment. J Allergy Clin Immunol. 2004 Sep;114(3):465-74; quiz 475. doi: 10.1016/j.jaci.2004.02.049. PMID 15356542
- [Background] Kaplan AP. What the first 10,000 patients with chronic urticaria have taught me: a personal journey. J Allergy Clin Immunol. 2009 Mar;123(3):713-7. doi: 10.1016/j.jaci.2008.10.050. Epub 2008 Dec 10. No abstract available. PMID 19081615
- [Background] Staevska M, Popov TA, Kralimarkova T, Lazarova C, Kraeva S, Popova D, Church DS, Dimitrov V, Church MK. The effectiveness of levocetirizine and desloratadine in up to 4 times conventional doses in difficult-to-treat urticaria. J Allergy Clin Immunol. 2010 Mar;125(3):676-82. doi: 10.1016/j.jaci.2009.11.047. PMID 20226302